CLINICAL TRIAL: NCT02569177
Title: Evaluation of the Association Between Heart Type Fatty-acid Binding Proteins and High Sensitive Troponin and Postoperative Myocardial Infarction in Patients Undergoing Cardiac Surgery.
Brief Title: Biomarkers for Postoperative Myocardial Infarction in Cardiac Surgery.
Status: Withdrawn | Type: Observational
Why Stopped: Due to lack of funding
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Dr. B. van Zaane, MD, PhD, UMC Utrecht
Other Study IDs: NL46363.041.14
Record Dates: First submitted 2015-09-28; First posted 2015-10-06 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Myocardial Infarction
Keywords: myocardial infarction; cardiac surgery; troponin; heart-type fatty acid binding protein
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be drawn before incision (baseline), during cardiopulmonary bypass and after release of the aortic cross clamp. Subsequently, blood samples will be drawn on arrival at the intensive care unit and three and six hours after arrival. On post-operative day 1 and 2 blood samples will be drawn on the ICU or the medium care. All samples will be stored according the hospital blood banking protocol and analyzed at once at the end of the study. Left over material will be discarded after all necessary analysis has been conducted.
Oversight: Data Monitoring Committee: No

SUMMARY:
Myocardial infarction and subsequent myocardial injury after cardiac surgery occurs in 7-15% of patients undergoing cardiac surgery and is associated with an increased length of stay, and reduced short- and long-term survival. Cardiac troponin is considered to be a cornerstone in the diagnosis of a myocardial infarction. Heart-type Fatty Acid-Binding Protein (H-FABP) is a new sensitive biomarker for myocardial injury. The effectiveness of using the combination of H-FABP with Troponin to diagnose myocardial injury within 6 hours after the onset of ischemia is well reported. Previous studies in non-surgical patients have associated increased H-FABP with an increased risk of subsequent death and major cardiac events. The prognostic value in cardiac surgery patients has not been studied extensively.

The objective is to estimate the association between biomarkers of myocardial injury and myocardial infarction in patients undergoing cardiac surgery. Myocardial infarction will be established with both a new and very early marker of myocardial injury (Heart-type Fatty Acid Binding Proteins) as well as to a known early marker of such injury (Cardiac troponin).

DETAILED DESCRIPTION:
Specific aims:

1. To obtain an estimate of the association between a new very early marker of postoperative myocardial injury H-FABP and postoperative myocardial infarction.
2. To obtain an estimate of the association between cTn-I and postoperative myocardial infarction.
3. To obtain an estimate of the correlation between H-FABP elevation and cTn-I elevation in patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* isolated coronary artery bypass grafting
* isolated valve surgery
* combined coronary artery bypass grafting and valve surgery

Exclusion Criteria:

* emergency surgery patients
* (suspected) sepsis
* pulmonary embolism
* renal failure (Glomerular filtration rate < 40 ml/min)
* off pump cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Postoperative myocardial infarction | 30 days after cardiac surgery
  The occurence of postoperative myocardial infarction is imported from the Board Heart interventions Netherlands registry (BHN registry). For every patient undergoing cardiac surgery in the UMCU the cardiothoracic department determines whether the patient had a postoperative myocardial infarction or not and fills out the related information in the BHN registry.

SECONDARY OUTCOMES:
Mortality | 30-days and 1-year after cardiac surgery
Hospital length of stay | 1 year after cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Bas van Zaane, Md, PhD, Principal Investigator — UMC Utrecht

REFERENCES:
- [Background] Domanski MJ, Mahaffey K, Hasselblad V, Brener SJ, Smith PK, Hillis G, Engoren M, Alexander JH, Levy JH, Chaitman BR, Broderick S, Mack MJ, Pieper KS, Farkouh ME. Association of myocardial enzyme elevation and survival following coronary artery bypass graft surgery. JAMA. 2011 Feb 9;305(6):585-91. doi: 10.1001/jama.2011.99. PMID 21304084
- [Background] Yau JM, Alexander JH, Hafley G, Mahaffey KW, Mack MJ, Kouchoukos N, Goyal A, Peterson ED, Gibson CM, Califf RM, Harrington RA, Ferguson TB; PREVENT IV Investigators. Impact of perioperative myocardial infarction on angiographic and clinical outcomes following coronary artery bypass grafting (from PRoject of Ex-vivo Vein graft ENgineering via Transfection [PREVENT] IV). Am J Cardiol. 2008 Sep 1;102(5):546-51. doi: 10.1016/j.amjcard.2008.04.069. Epub 2008 Jul 2. PMID 18721510
- [Background] Muehlschlegel JD, Perry TE, Liu KY, Fox AA, Collard CD, Shernan SK, Body SC. Heart-type fatty acid binding protein is an independent predictor of death and ventricular dysfunction after coronary artery bypass graft surgery. Anesth Analg. 2010 Nov;111(5):1101-9. doi: 10.1213/ANE.0b013e3181dd9516. Epub 2010 May 10. PMID 20457766